CLINICAL TRIAL: NCT06072794
Title: A Proof of Concept Study to Evaluate Exosomes From Human Mesenchymal Stem Cells in Women With Premature Ovarian Insufficiency (POI)
Acronym: VL-POI-01
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Vitti Labs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VL-POI-01
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Premature Ovarian Insufficiency; Diminished Ovarian Reserve
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a dose escalation study. The study participants are organized in groups of 3 where each participant will receive one study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: VL-PX10

INTERVENTIONS:
Drug: VL-PX10 — VL-PX10 is a decellularized product consisting of proteins, lipids, and nucleic acids derived from human placenta mesenchymal stem cells.

SUMMARY:
The VL-POI-01 study is designed to evaluate the safety and efficacy of human placental mesenchymal stem cell derived exosome treatment in patients with premature ovarian insufficiency (POI) and diminished ovarian reserve.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) is a devastating disease for young women who have not yet completed childbearing. The prevalence of this condition is on the rise due to the increasing number of cancer survivors and the delay in childbearing age. Current treatment options available are very limited. Stem cell therapy has been shown to be beneficial and effective in various disease processes and the safety has been assessed in multiple clinical trials. The regenerative potential of mesenchymal stem cells is increasingly attributed to the paracrine effects of exosomes. Exosomes consist of bioactive lipids, nucleic acids, and proteins which play a key role in intercellular communication. Exosome therapy is considered a safe and effective therapy since it offers a cell-free approach. VL-PX10 is a decellularized exosome product derived from human placental derived mesenchymal stem cells.

This interventional pilot study will investigate the ability of intravenous injection of VL-PX10 to restore steroidogenesis, folliculogenesis, and support quality of life improvement, resumption of menstruation, and reversal of infertility in patients with POI and diminished ovarian reserve.

This is an open label study. All patients entering this study will be treated with VL-PX10. Participant duration will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and communicate in English language
* Female of age 18-43 years
* Diagnosis of premature ovarian insufficiency based on ESHRE Guidelines (i) oligo/amenorrhea for at least 4 months, and (ii) an elevated FSH level >25 IU/L on two occasions >4 weeks apart, or diagnosis of low ovarian reserve defined as: Basal FSH value >10 IU/L or failure of prior attempts of assisted reproductive techniques due to limited ovarian response (poor responders)
* Normal karyotype 46, XX, and no known history FMR1 premutation (fragile X syndrome)
* Baseline AMH levels ≤ 1.0 ng/mL
* Presence of at least one ovary
* Normal uterine anatomy (by any clinically and/or imaging acceptable methods)
* Normal thyroid function as evident by normal serum Thyroid Stimulating Hormone (TSH) levels
* For subjects who had contraception before, the duration of amenorrhea should be more than 3 months after discontinuation of the oral contraception pill (OCP) or more than 6 months after discontinuation of Depo Provera (or similar) therapies
* Agree to report any pregnancy to the research staff immediately
* Willing and able to comply with study requirements and follow up instructions
* Patient with known history of endometriosis or polycystic ovarian syndrome
* If subject is planning to pursue pregnancy: presence of at least unilateral tubal patency (with any clinically acceptable methods)

Exclusion Criteria:

* Currently pregnant or breast-feeding
* Has a history of, or evidence of current gynecologic malignancy, breast cancer or other estrogen responsive cancer or any other malignancy within the past five years
* Subjects with FMR1 premutation (fragile X syndrome), a BMP15 mutation or family history of a first degree relative with POI
* Presence of adnexal masses indicating the need for further evaluation
* Major mental health disorder that precludes participation in the study
* Active substance abuse or dependence
* Current or recent (within the past 2 weeks) use of the following medications: Oral or systemic corticosteroids, Hormones (estrogen, progestin, oral contraceptives), Danazol, anticoagulants, herbal or botanical supplements with possible hormonal effects. Washout will be allowed (2 weeks from screening)
* Subjects under hormonal treatments including hormone replacement therapy (HRT) for osteoporosis, cardiovascular disease, or recalcitrant vasomotor symptomatology within 3 months from screening
* Subjects with a history of breast cancer or other estrogen responsive cancer within 5 years from screening
* Subjects with existing malignant neoplasm, under active management for malignant neoplasm or under active surveillance for malignant neoplasm within 5 years from screening
* Subjects with history of thromboembolic events such as pulmonary embolism, stroke, or ischemic heart disease
* Subjects with uncontrolled hypertension, kidney disease, liver disease, or polycystic ovary syndrome (PCOS) as defined below:

  * Uncontrolled hypertension: Systolic BP ≥ 140 and/or Diastolic BP ≥90 in patients taking anti-hypertensive treatment
  * Kidney Disease: an estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m^2 (Incase the result is above/below acceptable range, one repeat test is acceptable)
  * Liver Disease: Serum aminotransferase (ALT or AST) levels > 2x ULN
  * PCOS criteria: Oligo-anovulation (Irregular periods), antral follicle count (AFC) >12 measuring 2-9mm, hyperandrogenism (elevated testosterone and DHEA levels), clinical hirsutism
* Subjects with untreated endocrinopathies including Cushing's disease, thyroid disease, congenital adrenal hyperplasia and hyperprolactinemia
* Subjects with intra-uterine devices (IUDs)
* Subjects who are allergic to low-molecular-weight heparin sodium or human albumin
* Medical conditions that are contraindicated in pregnancy
* Type I or Type II diabetes mellitus, or if receiving antidiabetic medications within 3 months from screening
* Known anemia (Hemoglobin < 11 g/dL)
* History of deep venous thrombosis, and/or pulmonary embolus
* History of cerebrovascular disease
* History of contrast media allergy
* Known heart disease (New York Heart Association Class II or higher)
* Known Liver disease (defined as Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >2 times normal, or total bilirubin >2.5mg/dL)
* Known Renal disease (defined as Blood urea nitrogen (BUN) >30 mg/dL or serum creatinine > 1.6 mg/dL)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with premature ovarian insufficiency
Enrollment: 9 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  The number of treatment-emergent adverse events.

SECONDARY OUTCOMES:
Follicle Stimulating Hormone Levels | 2 years
  50% reduction in follicle stimulating hormone values.
Anti-Müllerian Hormone Levels | 2 years
  30% increase in anti-Müllerian hormone levels.
Estradiol Levels | 2 years
  30% increase in estradiol levels.
Antral Follicle Counts | 2 years
  Increased antral follicle counts.

CONTACTS AND LOCATIONS:
Locations (1):
- Optimal Health Associates, Oklahoma City, Oklahoma, United States